CLINICAL TRIAL: NCT06439329
Title: STOP (Shared Decision Making to Treat Or Prevent) HIV in Justice Populations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000037052; 1R61DA060625-01 (NIH)
Record Dates: First submitted 2024-05-28; First posted 2024-06-03 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Substance Use Disorders
MeSH Terms: conditions — Substance-Related Disorders | interventions — Patient Freedom of Choice Laws

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Patient Navigation (PN) (Active Comparator): PNs are "near-peer" professionals who have shared lived experiences with participants and help them overcome barriers to accessing and engaging in quality care. PNs are trained and linked to PrEP/ART and SUD services. This manualized PN approach provides appointment scheduling to brick and mortar services only, and not to MHU or telehealth services.
  Interventions: Behavioral: Standard PN
- PN + Patient Choice (PC) (PN+PC) (Experimental): PNs working in the PN + PC arm will be trained to engage participants in selecting from the menu of options developed in the pilot. This menu of SUD and HIV prevention and treatment service delivery options will be created through bolstering and working with our CAB.
  Interventions: Behavioral: Standard PN; Behavioral: Patient Choice

INTERVENTIONS:
Behavioral: Standard PN — Standard of care
Behavioral: Patient Choice — Participants can select from a menu of options including brick and mortar services, Mobile Health Unit (MHU) or telehealth services.
  Arms: PN + Patient Choice (PC) (PN+PC)

SUMMARY:
This study seeks to compare the effectiveness of two Patient Navigation models of care to evaluate the proportion who initiate PrEP/ART and substance use/substance use disorder (SU/SUD) treatment. A standardized Patient Navigation (PN) arm will be compared with a shared decision-making model in the form of Patient Choice (PC) through the offer of a menu of existing community-based health service delivery options. This design will offer providers, correctional and public health authorities, payers and policy makers' timely and relevant data to assess the effectiveness of Patient Navigation and Patient Choice models of care as potentially useful re-entry and relapse prevention treatment options.

DETAILED DESCRIPTION:
This study will be done in two phases. Phase 1 the R61 portion of the project will be a Pilot Study, and Phase 2 the R33 portion of the project will be a Randomized Controlled Trail informed by the pilot.

The focus of this registration is the pilot study. In Year 1 (R61; Aim 1) the intervention of the patient choice menu of options of PrEP/ART and SUD treatment services for justice involved people who use drugs (PWUD) to supplement established peer navigation (PN +PC) will be developed and pilot tested in Western Connecticut only (Fairfield, Litchfield, Southern New Haven Counties).

Implementation procedures for this study include needs assessment survey and focus groups consisting of CAB members and PNs to assess the types of services available in their community, as well as gaps in services and ideas of how services can be improved. These needs assessment surveys and focus groups will occur 3 times throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* able to provide written informed consent in English or Spanish;
* living in the community of Western, CT, Dallas and Tarrant Counties in TX and Madison County, KY (potential for Fayette county as well);
* Those with current justice involvement (with in the past 6 months) (e.g., prison, jail, community supervision);
* willing to have HIV testing to determine negative or positive status;
* persons with HIV who report not currently taking ART and have a viral load >200 copies/mL in past 6 months OR persons who test negative for HIV who report not taking PrEP that meet CDC PrEP eligibility criteria in past 6 months, including (i) condomless sexual intercourse; and/or (ii) sharing IDU equipment with HIV positive or unknown status partner; and/or (iii) bacterial STI and;
* Having a history of opioid and/or stimulant use within 12 months prior to being in a controlled setting and/or in the last 6 months within the community

Implementation portion/CAB members:

* able to provide written informed consent in English or Spanish;
* working with persons with a history of justice involvement and substance use in the areas targeted for this project

PN Participants:

* able to provide written informed consent in English or Spanish;
* be employed at a project research site as a Patient Navigator

Exclusion Criteria:

* severe medical or psychiatric disability making participation unsafe;
* unable to provide consent.
* persons self-reporting pregnancy

Implementation portion/CAB members:

* persons self-reporting pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2024-10-03 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Feasibility/acceptability will be assessed using the CAB Community Needs Assessment | 3 months
  Attitudes toward acceptability and feasibility of the PN and PN+PC menu of options will be surveyed from CAB members using the needs assessment created during project ACTION as a foundation.
Feasibility/acceptability will be assessed using the Organizational Readiness for Implementing Change (ORIC) from the JCOIN Common Measure survey | 3 months
  Organizational readiness for implementing change (ORIC) will be surveyed at start of preparation and sustainment phases with CAB members to evaluate confidence and commitment to using the PN+PC approach.
Participant attitudes toward the interventions will be assessed using the Scales for Participant Alliance with Recovery Coach (SPARC) | 3 months
  Participant attitudes toward the PN and PN+PC implementation approach (rapport, satisfaction, linkage to services, engagement) will be collected at 3 months using the Scales for Participant Alliance with Recovery Coach; SPARC. The SPARC is scored on a Likert scale (1 = strongly disagree to 5 = strongly agree), higher scores indicate a high perception of the recovery coach alliance. There are six domains (engagement, satisfaction, rapport, motivation and encouragement, role model, and community linkage), and each domain score is between 10 and 50.
Percentage of participants with access to PrEP/ART services | 3 months
  Utilization of Services and PN Engagement data will be used to assess the percentage of participants with access to PrEP/ART services.
Percentage of participants with receipt of treatment | 3 months
  Defined as participants that have received a prescription for PrEP/ART

SECONDARY OUTCOMES:
Substance use treatment | 3 months
  Percentage of participants engaged in substance use disorder (SUD) treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Springer, MD, Principal Investigator — Yale University
Locations (1):
- 135 College St., Suite 280, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No